CLINICAL TRIAL: NCT07053605
Title: Clinical Study on Laparoscopic Resection of Splenic Artery Aneurysm With Preservation of Spleen
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Guo-Qing Jiang, Clinical Professor, Northern Jiangsu People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YZUC-013
Record Dates: First submitted 2025-06-23; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Splenic Artery Aneurysm; Immune Function; Hemodynamics
Keywords: Laparoscopy; resection of splenic artery aneurysm; Immune function; Hemodynamics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The laparoscopic resection of splenic artery aneurysm is performed by the same surgical team. (Experimental): The laparoscopic resection of splenic artery aneurysm with preservation of spleen is performed by the same surgical team.
  Interventions: Procedure: laparoscopic resection of splenic artery aneurysm with preservation of spleen

INTERVENTIONS:
Procedure: laparoscopic resection of splenic artery aneurysm with preservation of spleen — The laparoscopic resection of splenic artery aneurysm with preservation of spleen is performed by the same surgical team.

SUMMARY:
In this study, researchers examined the changes in related indicators such as immune function, splenic vein,proper hepatic artery, and portal venous hemodynamics following laparoscopic resection of a splenic artery aneurysm. We determined the changes in these patient-related indicators after surgical treatment and whether these changes could improve patient outcomes.

DETAILED DESCRIPTION:
Patients with Splenic Artery Aneurysm were recruited in accordance with the research inclusion criteria, and their general demographic information was collected. After thorough preoperative preparation, the same surgical team performed laparoscopic resection of the splenic artery aneurysm. Postoperatively,the same nursing team provided standardized care. Subsequently, patients received a standardized postoperative treatment protocol, which included pharmacotherapy, additional therapeutic interventions, and follow-up visits. During the treatment period, routine blood tests,liver function tests, coagulation function,immune function, as well as the hemodynamics of the portal vein, proper hepatic artery, and splenic vein were monitored preoperatively and at 7 days, 1 month, 3 months, 6 months, and 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic splenic artery aneurysms with a diameter>2 cm,ruptured splenic artery aneurysms,and splenic artery aneurysms with a diameter increase>0.5 cm/year.

Aneurysm located in the main trunk of the splenic artery. Informed consent to participate in the study.

Exclusion Criteria:

* Patients with malignancies Hepatic cirrhosis with portal hypertension peptic ulcer disease Recent peptic ulcer disease History of Hemorrhagic stroke Pregnancy hematological diseases Uncontrolled Hypertension Human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The immune function at 7 days after surgery | 7 days
  The level of the immune function(Complement C3; Complement C4; IgG; IgA; IgM;CD19;CD20;CD16;CD56;CD3;CD4) at 7 days after surgery.
The immune function at 1 month after surgery | 1 month
  The level of the immune function(Complement C3; Complement C4; IgG; IgA; IgM;CD19;CD20;CD16;CD56;CD3;CD4) at 1 month after surgery.
The immune function at 3 months after surgery | 3 months
  The level of the immune function(Complement C3; Complement C4; IgG; IgA; IgM;CD19;CD20;CD16;CD56;CD3;CD4) at 3 months after surgery.
The immune function at 6 months after surgery | 6 months
  The level of the immune function(Complement C3; Complement C4; IgG; IgA; IgM;CD19;CD20;CD16;CD56;CD3;CD4) at 6 months after surgery.
The immune function at 12months after surgery | 12months
  The level of the immune function(Complement C3; Complement C4; IgG; IgA; IgM;CD19;CD20;CD16;CD56;CD3;CD4) at 12months after surgery.
Routine blood tests (Erythrocyte Count; Hemoglobins; Red Cell Distribution Width; White Blood Cell Count; Neutrophils; Lymphocytes; Monocytes; Eosinophils; Basophils; Platelet Count; Mean Platelet Volume; Blood Platelet) at 1 month postoperatively. | 1 month
  1 month
Routine blood tests (Erythrocyte Count; Hemoglobins; Red Cell Distribution Width; White Blood Cell Count; Neutrophils; Lymphocytes; Monocytes; Eosinophils; Basophils; Platelet Count; Mean Platelet Volume; Blood Platelet) at 3 months postoperatively. | 3 months
  3 months
Routine blood tests (Erythrocyte Count; Hemoglobins; Red Cell Distribution Width; White Blood Cell Count; Neutrophils; Lymphocytes; Monocytes; Eosinophils; Basophils; Platelet Count; Mean Platelet Volume; Blood Platelet) at 6 months postoperatively. | 6 months
  6 months
Routine blood tests (Erythrocyte Count; Hemoglobins; Red Cell Distribution Width; White Blood Cell Count; Neutrophils; Lymphocytes; Monocytes; Eosinophils; Basophils; Platelet Count; Mean Platelet Volume; Blood Platelet) at 12 months postoperatively. | 12 months
  12 months
Hemodynamics (Vascular Diameter; Blood Flow Velocity) of the splenic vein,proper hepatic artery,and portal vein at 1 month postoperatively. | 1 month
  1 month
Hemodynamics (Vascular Diameter; Blood Flow Velocity) of the splenic vein,proper hepatic artery,and portal vein at 3 months postoperatively. | 3 months
  3 months
Hemodynamics (Vascular Diameter; Blood Flow Velocity) of the splenic vein,proper hepatic artery,and portal vein at 6 months postoperatively. | 6 months
  6 months
Hemodynamics (Vascular Diameter; Blood Flow Velocity) of the splenic vein,proper hepatic artery,and portal vein at 12 months postoperatively. | 12 months
  12 months
Thrombosis in the Portal Venous System. | 1 month
  1 month
Thrombosis in the Portal Venous System. | 3 months
  3 months
Thrombosis in the Portal Venous System. | 6 months
  6 months
Thrombosis in the Portal Venous System. | 12 months
  12 months

CONTACTS AND LOCATIONS:
Overall Officials: Guo-Qing Jiang, Study Chair — Clinical Medical College, Yangzhou University
Locations (1):
- Clinical Medical College, Yangzhou University, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No